CLINICAL TRIAL: NCT03379181
Title: Thermogenesis in Hyperthyroidism and Effect of Anti-Adrenergic Therapy
Acronym: HEAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EKNZ 2017-02044
Record Dates: First submitted 2017-12-07; First posted 2017-12-20 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Hyperthyroidism
Keywords: Brown adipose tissue (BAT); Hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Propranolol 80 mg (Experimental): Patients receive a single dose of 80 mg propranolol p.o.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Patients receive a single dose of 80 mg propranolol p.o.
  Other Names: beta blockade

SUMMARY:
The overall objective of the HEAT study is to determine the acute effect of propranolol on energy expenditure in patients suffering from hyperthyroidism and to evaluate the consequences of the change of hyper- to euthyroidism on metabolism during the course of treatment, especially with regard to the reaction to cold ambient temperatures.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Age 18 to 70 years
* Hyperthyroidism: Thyroid-stimulating Hormone (TSH) below 0.2 mU and free T4 at or above 25 pmol/L or free T3 at or above 8 pmol/L.

Exclusion Criteria:

* Contraindications to propranolol: hypersensitivity or allergy
* Therapy with a beta blocker for reasons other than hyperthyroidism (e.g. cardiac arrhythmia or heart failure)
* Treatment with amiodarone
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* History of asthma or chronic obstructive pulmonary disease
* Occlusive peripheral artery disease; Raynaud's syndrome.
* Other clinically significant concomitant disease states:

  * Known renal failure (GFR < 50 ml/min)
  * Known hepatic dysfunction
  * known heart failure or unstable angina pectoris
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons.
* ECG-criteria

  * Resting heart rate below 60 bpm
  * Complete left bundle branch block
  * Atrioventricular block (AV-block) grade 2 or 3

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
acute effect of propranolol on energy expenditure in patients suffering from hyperthyroidism | 90 minutes after propranolol application
  difference in resting energy expenditure (REE) measured single 90 minutes after an oral dose of 80 mg of propranolol compared to resting energy expenditure measured during the thirty minutes prior to administration of propranolol (ΔREEPropranolol).

SECONDARY OUTCOMES:
Respiratory quotient (RQ) before and after administration of propranolol. | 90 minutes after propranolol application
  Difference in respiratory quotient (RQ) before and after administration of propranolol.
Difference in skin temperature | 90 minutes after propranolol application
  Supraclavicular skin temperature in patients with hyperthyroidism after a single dose of 80 mg Propranolol compared to supraclavicular temperature before Propranolol.
Difference in REE from hyperthyroid to euthyroid state | after 3 to 4 months
  indirect calorimetry to determine resting energy expenditure
Difference in REE hyperthyroid state to euthyroid state | after 6 to 7 months
  indirect calorimetry to determine resting energy expenditure
Change in Body composition: percent body fat | after 3 to 4 months
  dual xray absorption scan
Cold induced thermogenesis (CIT) in patients with hyperthyroidism | after 3 to 4 months
  Cold induced thermogenesis: Increase in energy expenditure above resting metabolic rate in response to a mild cold stimulus during hyperthyroidism as compared to euthyroidism.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias J Betz, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Department of Endocrinology, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Senn JR, Loliger RC, Fischer JGW, Bur F, Maushart CI, Betz MJ. Acute effect of propranolol on resting energy expenditure in hyperthyroid patients. Front Endocrinol (Lausanne). 2023 Jan 19;13:1026998. doi: 10.3389/fendo.2022.1026998. eCollection 2022. PMID 36743920
- [Derived] Maushart CI, Senn JR, Loeliger RC, Siegenthaler J, Bur F, Fischer JGW, Betz MJ. Resting Energy Expenditure and Cold-induced Thermogenesis in Patients With Overt Hyperthyroidism. J Clin Endocrinol Metab. 2022 Jan 18;107(2):450-461. doi: 10.1210/clinem/dgab706. PMID 34570185